CLINICAL TRIAL: NCT00804804
Title: Aging,Sleep and Cognitive Process
Brief Title: Aging, Sleep, Cognitive Process
Acronym: SOMVIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean Pierre LEROY/ Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2008/17
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: BIOLOGICAL CLOCKS
Keywords: Sleep; aging; cognitives processes; constant routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Y1 (Experimental): young volunteers (20-30 years), morningness chronotype
  Interventions: Other: Sleep deprivation and multiple rest
- Y2 (Experimental): young volunteers (20-30 years), eveningness chronotype
  Interventions: Other: Sleep deprivation and multiple rest
- O1 (Experimental): Aged volunteers (65-75 years), morningness chronotype
  Interventions: Other: Sleep deprivation and multiple rest
- O 2 (Experimental): aged volunteers (65-75 years), eveningness chronotype
  Interventions: Other: Sleep deprivation and multiple rest

INTERVENTIONS:
Other: Sleep deprivation and multiple rest — To determine the evolution of the executive functions during a 40-hour extended wakefulness period or during a 40-hour multiple nap protocol in constant experimental conditions of confinement
  Arms: Y1
Other: Sleep deprivation and multiple rest — To determine the evolution of the executive functions during a 40-hour extended wakefulness period or during a 40-hour multiple nap protocol in constant experimental conditions of confinement
  Arms: Y2
Other: Sleep deprivation and multiple rest — To determine the evolution of the executive functions during a 40-hour extended wakefulness period or during a 40-hour multiple nap protocol in constant experimental conditions of confinement
  Arms: O1
Other: Sleep deprivation and multiple rest — To determine the evolution of the executive functions during a 40-hour extended wakefulness period or during a 40-hour multiple nap protocol in constant experimental conditions of confinement
  Arms: O 2

SUMMARY:
The aim of the study is to determine the impact of aging, circadian rhythms and sleep deprivation on executive performances. Volunteers will complete a 40-hour extended wakefulness period in constant condition (semi-recumbent posture in bed, constant dim light levels < 10 lux, food and liquid intake at regular intervals) in order to control the circadian system. The volunteers will not be allowed to sleep in the sleep deprivation protocol ("high sleep pressure protocol") and will adopt a short wakefulness/sleep cycle (150/75 minutes) in the multiple nap protocol ("low sleep pressure protocol"). Tests and scales will be repeated every 3H45

DETAILED DESCRIPTION:
Social evolutions (nocturnal activity, shift work) have consequently reduced average sleep duration average. In addition, aging leads to a physiological reduction of nocturnal sleep duration.

Many studies have shown that extended wakefulness impairs nocturnal performances measured with a simple reaction time test (SRTT) and that this decrement is also age-related. In deed, young subjects (20-30 years) are more affected than old subjects (50-60 years) during an extended wakefulness period.

The results obtained in confinement constant conditions, associated to a high or low sleep pressure, show that this difference observed between young and old subjects should be essentially related to a reduced circadian regulation (ex : reduced melatonin secretion) with age rather than to a reduced sleep pressure (homeostatic regulation) as previously suggested. However, studies on confinement have shown that sleep pressure (identified during the sleep period with the EEG delta band) could be reduced with aging specifically on the anterior brain regions (frontal regions).

It is well-known that executive performances (related to frontal lobes functioning) are affected by extended wakefulness, but respective effects of age, circadian system and sleep pressure in this decrement remain unknown.

The aim of this study is to determine the evolution of the executive functions during a 40-hour extended wakefulness period ("high sleep pressure protocol") or during a multiple nap protocol ("low sleep pressure protocol") according to the subjects' age, in constant experimental conditions of confinement.

It's a repeated measurements study with protocol (sleep deprivation and multiple naps) and time of day as within factors and age group (young versus older subjects) as between factor

ELIGIBILITY:
Inclusion Criteria:

* excessive daytime sleepiness (Epworth Sleepiness Scale score > 9),
* sleep complaint such as sleep apnea or insomnia (Basic Nordic Sleep Questionnaire, items score < 4 except questions 3, 4 and 15a for aged volunteers),
* not intermediate in terms of morningness and eveningness according to the Horne-Ostberg questionnaire for young volunteers
* absence of psychopathology evidenced during psychologist interview or on the Symptom Check List (SCL-90R score>59)
* sleep efficiency evidenced by actimetry (>85%) during 7 days
* absence of apnea/hypopnea syndrome (RDI<15)
* absence of periodic movement disorder (MPS<15)
* regular sleep schedule during 3 days before study participation
* affiliated to the french health care system

Exclusion Criteria:

* volunteers with sleep disorders or organic disorders affecting sleep,
* poor sleep hygiene or abnormal usual sleep patterns,
* night workers or shift-workers,
* substance abusers (caffeine, drug, or alcohol).

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Executive functions will be evaluated by a Go/NoGo task and a Stop Signal. Performances will be measured with a visual simple reaction time task | every 3h45

SECONDARY OUTCOMES:
Nocturnal sleep quality before and after 2 constant conditions measured by PSG Sleep pressure quantified by Karolinska test and EEG delta band Subjective sleepiness and fatigue evaluated by Karolinska sleepiness scale and visual analogue scale | every 3h45

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PHILIP, MD,PHD, Principal Investigator — University Hospital Bordeaux France
Locations (3):
- France (3):
  - Genpphass, Bordeaux
  - Uh Purpan, Toulouse
  - Medes-Imps, Toulouse